CLINICAL TRIAL: NCT01929655
Title: A Single-arm, Open-label, Multicenter, Phase II Study of BAY88-8223 in the Treatment of Japanese Patients With Symptomatic Castration-resistant Prostate Cancer (CRPC) With Bone Metastases
Brief Title: Japanese BAY88-8223 Monotherapy Phase II Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16430
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Prostatic Neoplasms
Keywords: Phase II; symptomatic castration-resistant prostate cancer; bone metastases
MeSH Terms: conditions — Prostatic Neoplasms | interventions — radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radium-223 dichloride (Experimental)
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — BAY88-8223, 50 kBq/kg will be administered as slow bolus intravenous injection 6 times at intervals of 4 weeks between each administration

SUMMARY:
To evaluate the efficacy and safety of the best standard of care plus BAY88-8223 in Japanese patients with CRPC and bone metastases after a multiple administration

ELIGIBILITY:
Inclusion Criteria:

* Have received docetaxel or not eligible for the first course of docetaxel, i.e. patients who are not fit enough and willing.
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Multiple bone metastases
* Either regular (not occasional) analgesic medication use for cancer-related bone pain or treatment with external beam radiotherapy (EBRT) for bone pain.
* Best standard of care(BSoC) is regarded as the routine standard of care.

Exclusion Criteria :

* Treatment with cytotoxic chemotherapy within previous 4 weeks, or planned during the treatment period
* History of visceral metastasis, or presence of visceral metastasis

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Percentage of change in total alkaline phosphatase from baseline at 12 weeks | Baseline and 12 weeks

SECONDARY OUTCOMES:
Percentage of change in total alkaline phosphatase at the end of treatment | Baseline and 24 weeks
Percentages of change in bone ALP at 12 weeks | Baseline and 12 weeks
Percentages of change in bone ALP at the end of treatment | Baseline and 24 weeks
The proportion of subjects who have total alkaline phosphatase normalization at 12 weeks | 12 weeks
The proportion of subjects who have total alkaline phosphatase normalization at the end of treatment | 24 weeks
The proportion of subjects who have bone alkaline phosphatase normalization at 12 weeks | 12 weeks
The proportion of subjects who have bone alkaline phosphatase normalization at the end of treatment | 24 weeks
Time to prostate specific antigen progression | 24 weeks
Overall survival | 3 years
Percentages of change in biomarkers of bone turnover at each time point | Baseline and 36 weeks
Number of participants with drug related adverse events and serious adverse events as a measure of safety and tolerability | 3 years
Incidence of treatment-emergent adverse events (TEAEs) | 24 weeks plus 30 days
Number of participants with abnormal laboratory values | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (14):
- Japan (14):
  - Kashiwa, Chiba
  - Sapporo, Hokkaido
  - Kanazawa, Ishikawa-ken
  - Yokohama, Kanagawa
  - Sendai, Miyagi
  - Sayama, Osaka
  - Hamamatsu, Shizuoka
  - Bunkyo-ku, Tokyo
  - Koto-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Chiba
  - Fukuoka
  - Kumamoto
  - Okayama

REFERENCES:
- [Derived] Matsubara N, Nagamori S, Wakumoto Y, Uemura H, Kimura G, Yokomizo A, Kikukawa H, Mizokami A, Kosaka T, Masumori N, Kawasaki Y, Yonese J, Nasu Y, Fukasawa S, Sugiyama T, Kinuya S, Hosono M, Yamaguchi I, Tsutsui H, Uemura H. Phase II study of radium-223 dichloride in Japanese patients with symptomatic castration-resistant prostate cancer. Int J Clin Oncol. 2018 Feb;23(1):173-180. doi: 10.1007/s10147-017-1176-0. Epub 2017 Aug 2. PMID 28770408